CLINICAL TRIAL: NCT01679821
Title: Prevalence of Signs and Symptoms of Temporomandibular Disorders (TMD) in Patients Wearing Double Complete Dentures, Removable Partial Dentures and Dentistry Students at State University of West of Paraná - UNIOESTE
Brief Title: Prevalence of Signs and Symptoms of TMD in Patients Wearing Double Complete Dentures, RPD and in Dentistry Students.
Status: Completed | Type: Observational
Sponsor: Universidade Estadual do Oeste do Paraná (Other)
Responsible Party: Principal Investigator, Maristela Maria Galina Pezzini, Associate Professor, Department of Occlusion, State University of West of Paraná - UNIOESTE, Cascavel, PR, Brazil, Universidade Estadual do Oeste do Paraná
Other Study IDs: 538/2010-CEP
Record Dates: First submitted 2012-09-01; First posted 2012-09-06 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-09

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Temporomandibular disorders.; Dental prosthesis.; Dental students
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — The sample consisted of 210 individuals, aged 19-90 years (average 44.5 years) of both genders, divided into 3 groups:
  Group 1 - seventy dental students of State University of West of Paraná - UNIOESTE; Group 2 - seventy patients treated at the UNIOESTE Dental Clinic that wore removable partial denture (partially edentulous); Group 3 - seventy patients with double complete dentures treated in Center for Dental Specialties of Cascavel - PR.
  Students in orthodontic treatment or with less than one year after the end of orthodontic treatment were excluded from the research. Patients wearing a complete denture in one maxillary and a removable partial denture in another maxillary, and patients wearing just one complete denture were not included in the research.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Dental students: Seventy dental students of State University of West of Paraná - UNIOESTE. Students in orthodontic treatment or with less than one year after the end of orthodontic treatment were excluded from the research. A questionnaire and a clinical examination were employed.
  Interventions: Other: A questionnaire and a clinical examination
- Removable partial denture: Seventy patients treated at the UNIOESTE Dental Clinic that wore removable partial denture (partially edentulous). Patients wearing a complete denture in one maxillary and a removable partial denture in another maxillary were not included in the research. A questionnaire and a clinical examination were employed.
  Interventions: Other: A questionnaire and a clinical examination
- Double complete denture: Seventy patients with double complete dentures treated in Center for Dental Specialties of Cascavel, Paraná, Brazil. Patients wearing just one complete denture were not included in the research. A questionnaire and a clinical examination were employed.
  Interventions: Other: A questionnaire and a clinical examination

INTERVENTIONS:
Other: A questionnaire and a clinical examination — Seventy dental students of State University of West of Paraná - UNIOESTE, seventy patients treated at the UNIOESTE Dental Clinic that wore removable partial denture (partially edentulous) and seventy patients with double complete dentures treated in Center for Dental Specialties of Cascavel, Paraná, Brazil. Students in orthodontic treatment or with less than one year after the end of orthodontic treatment were excluded from the research. Patients wearing a complete denture in one maxillary and a removable partial denture in another maxillary, and patients wearing just one complete denture were not included in the research.

SUMMARY:
It was proposed in this study to evaluate the prevalence of TMD signs and symptoms in State University of West of Parana's dental students with natural dentition, in patients with removable partial dentures and double complete dentures.

DETAILED DESCRIPTION:
The Temporomandibular Disorder (TMD) has a high prevalence among the population. Objectives: To evaluate the prevalence of signs and symptoms of TMD. Methodology: 210 randomly selected individuals were evaluated, being divided into three groups with seventy individuals each: Group 1 - dental students with natural dentition. Group 2 - patients with removable partial dentures. And Group 3 - patients with double complete dentures. The questionnaire of the American Academy of Orofacial Pain for triage was employed, then, clinical evaluation was carried out.

ELIGIBILITY:
Inclusion Criteria:

- Patients wearing double complete denture, patients wearing just removable partial denture and dentate students.

Exclusion Criteria:

Students in orthodontic treatment or with less than one year after the end of orthodontic treatment were excluded from the research.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Seventy dental students of State University of West of Paraná - UNIOESTE, seventy patients treated at the UNIOESTE Dental Clinic that wore removable partial denture (partially edentulous) and seventy patients with double complete dentures treated in Center for Dental Specialties of Cascavel, Paraná, Brazil.
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2010-12; Primary Completion 2011-03 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Assessment of the prevalence of signs and symptoms of temporomandibular disorders in patients with removable partial dentures, complete double dentures and toothed. | 5 months

SECONDARY OUTCOMES:
questionnaire for selection of orofacial pain and temporomandibular disorders recommended by the American Academy of Orofacial Pain | 5 monts

OTHER OUTCOMES:
Clinical examination | 5 months
  A clinical examination, which was divided into parts, namely: identification and analysis; part of the Axis I of RDC/TMD - Research Criteria for Temporomandibular Disorders; muscle palpation; and for patients with dentures, the history and clinical evaluation of them

CONTACTS AND LOCATIONS:
Overall Officials: Maristela Pezzini, Professor, Principal Investigator — Universidade Estadual do Oeste do Paraná; Thaisa Bordin, Student, Principal Investigator — Universidade Estadual do Oeste do Paraná
Locations (1):
- Universidade Estadual do Oeste do Paraná, Cascavel, Paraná, Brazil